CLINICAL TRIAL: NCT04010552
Title: A Phase II Trial to Assess the Evolution of KRAS Mutation Load by Liquid Biopsy in Patients With Resectable Pancreatic Ductal Adenocarcinoma Treated With Neoadjuvant NALIRINOX
Brief Title: Nalirinox Neo-pancreas RAS Mut ctDNA Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundación de investigación HM (Other)
Collaborators: Syntax for Science, S.L (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FiHM006
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Resectable Pancreatic Ductal Adenocarcinoma

STUDY DESIGN:
Intervention Model Description: This study is a multicenter, single-arm, interventional, open-label, non-randomized, phase II clinical trial, to evaluate the association of KRAS mutational load and histological tumour response after chemotherapy treatment in patients with PDAC. Due to its single-arm design patients will be assigned to a single group (non-randomized) and there will be no masking (open-label).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NALIRINOX treatment (Experimental): Patients will be treated with NALIRINOX, a combination of three chemotherapy agents: 5- FU/LV, nal-IRI, and oxaliplatin. Treatment regimen will consist of 8 cycles of neoadjuvant NALIRINOX prior to surgery and trial duration is expected to be 24 months.
  Interventions: Drug: NALRINOX combination

INTERVENTIONS:
Drug: NALRINOX combination — NALRINOX: combination of three chemotherapy agents: 5- FU/LV, nal-IRI, and oxaliplatin

SUMMARY:
Pancreatic cancer has an unfavorable prognosis with a reduced possibility of long-term survival. The only treatment with curative potential is surgery, but it is only possible in 15-20% of cases.

There are patients with clear criteria for surgical entry, others at the limit of the possibility of surgery, and patients with such advanced disease (either locally or with metastasis) that surgery is not indicated.

The objective of neoadjuvant chemotherapy treatment (received before surgery) is to reduce the tumor before surgery and reduce the risk of subsequent metastases and local recurrences, in borderline tumors or those resectable with high-risk criteria.

The FOLFIRINOX scheme, composed of 5-fluorouracil / folinic acid, oxaliplatin and irinotecan, is recommended as neoadjuvant treatment, but the response is still low. This study will use a modified FOLFIRINOX (NALIRINOX) regimen with a form of irinotecan attached to liposomes that allows greater action on tumor cells.

Mutations in the KRAS gene are associated with a greater growth capacity of tumor cells and are present in 90% of pancreatic cancers in advanced stages. They would be less frequent in earlier phases but little is known about the impact that chemotherapy treatment and subsequent surgery could have on the increase or decrease of these mutations, as well as their implication. The follow-up of these mutations with repeated pancreatic biopsies is not viable, but it can be monitored by simple blood samples in which the genetic material of the tumor can be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or females, aged 18 years or older
2. Histologically or cytologically confirmed diagnosis of PDAC
3. Candidates for pancreatic cancer surgery (no comorbidities that can exclude for surgery)
4. Life expectance of at least 12 months
5. Carbohydrate antigen 19-9 (CA19-9) levels < 500 U/ml
6. ECOG performance status ≤ 1
7. Adequate bone marrow function:

   * Hemoglobin >9 g/dL
   * Platelets >100.000 µL
   * Absolute neutrophil count (ANC) >1500 µl
   * Serum albumin > 3 g/dL
8. Adequate hepatic function:

   * Aspartate aminotransferase (AST) <3 upper limits of normal (ULN)
   * Alanine Aminotransferase (ALT) <3 ULN
   * Total Bilirubin < 1.5 ULN. If values are > 1.5 external drainage with a stent is allowed.
9. Adequate renal function:

   - Clearance of creatinine (ClCr) >60 ml/min
10. Sexually active men and women of childbearing potential must use efficient contraceptive methods. Contraceptive methods comprise: oral contraceptives, intrauterine devices, sexual abstinence, tubal ligation, IUD, barrier methods or another contraceptive considered appropriate by the investigator. Women of childbearing potential must have a negative serum pregnancy test before study entry.
11. Agree to participate and signed the ICF.

Exclusion Criteria:

1. Patients with metastatic disease
2. Patients ≥ 75 years.
3. Uncontrolled coagulopathy
4. Patients with a contraindication to surgery (locally advanced disease or patients not amenable to pancreatic surgery due to a previous comorbidity)
5. Patients with prior or concurrent malignant disease that required treatment with chemotherapy in the past.
6. Previous cytotoxic therapy within 36 months for other no-cancer disease (ie arthritis rheumatoid)
7. Known or suspected reactions to any component of the study medication (5-FU/LV, nal- IRI or oxaliplatin) or to components of similar chemical or biologic composition
8. Concurrent participation in any other clinical trial likely to interfere with the therapeutic schedule
9. Human immunodeficiency virus (HIV) positivity, active Hepatitis B or Hepatitis C infection.
10. Uncontrolled illness including ongoing or active infection, symptomatic congestive heart failure, unstable angina, cardiac arrhythmia, myocardial infarction, or left ventricular ejection fraction (LVEF) < 50, among others, or psychiatric illness/social situations that would limit compliance with study requirements.
11. Pregnant or breast-feeding women.
12. Any medical condition that, based on investigator's criteria, places the subject at risk, makes the subject ineligible or may jeopardize protocol compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with a good histological tumour response in the resected specimens after neoadjuvant chemotherapy with NALIRINOX and surgical removal according to the Ryan's classification in KRAS positive and negative patients | 8 weeks after surgical intervention

SECONDARY OUTCOMES:
R0 resection | Through the study completion (estimated to be 15 months)
1-year survival and Overal survival (OS) in baseline KRAS+ and KRAS- subjects | Through the study completion (estimated to be 15 months)
Progression Free Survival (PFS) | Through the study completion (estimated to be 15 months)
Assessment of the proportion of KRAS- subjects switching to KRAS+ (and from KRAS+ to negative) after neoadjuvant NALIRINOX | Through the study completion (estimated to be 15 months)
Assessment of the number of KRAS- subjects switching to KRAS+ (and from KRAS+ to negative) after neoadjuvant NALIRINOX | Through the study completion (estimated to be 15 months)
Impact on R0 resection for KRAS- subjects switching to KRAS+ (and from KRAS+ to negative) after neoadjuvant NALIRINOX | Through the study completion (estimated to be 15 months)
Impact on histological tumour response for KRAS- subjects switching to KRAS+ (and from KRAS+ to negative) after neoadjuvant NALIRINOX | Through the study completion (estimated to be 15 months)
Impact on PFS for KRAS- subjects switching to KRAS+ (and from KRAS+ to negative) after neoadjuvant NALIRINOX | Through the study completion (estimated to be 15 months)
Impact on 1-year survival for KRAS- subjects switching to KRAS+ (and from KRAS+ to negative) after neoadjuvant NALIRINOX | Through the study completion (estimated to be 15 months)
Impact on OS for KRAS- subjects switching to KRAS+ (and from KRAS+ to negative) after neoadjuvant NALIRINOX | Through the study completion (estimated to be 15 months)
Number of AEs and SAEs (according to CTCAE) to describe the safety profile of the neoadjuvant NALIRINOX scheme | Through the study completion (estimated to be 15 months)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Cubillo, MD, Study Director — Director
Locations (3):
- Spain (3):
  - Hestia Duran I Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Madrid Sanchinarro, PAU de Sanchinarro, Madrid
  - Hospital Universitari Vall D'Hebron, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided